CLINICAL TRIAL: NCT07343960
Title: A Phase I, Single-dose, Non-randomized, Open-label, Parallel Group Study to Assess the Pharmacokinetics and Safety of Capivasertib in Participants With Moderate Hepatic Impairment
Brief Title: A Phase I Study to Investigate the Pharmacokinetics and Safety of Capivasertib in Participants With Moderate Hepatic Impairment
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D3615C00004
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Moderate Hepatic Impairment
Keywords: Hepatic function; Anti-cancer agent; Pyrrolopyrimidine-derived compound; Liver metabolism; Serine/threonine protein kinase AKT; Pharmacokinetics
MeSH Terms: interventions — capivasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test: Capivasertib in Moderate hepatic impairment (Experimental): Participants with moderate hepatic impairment will receive a single dose of capivasertib.
  Interventions: Drug: Capivasertib
- Control: Capivasertib in Normal hepatic function (Experimental): Participants with normal hepatic function will receive a single dose of capivasertib.
  Interventions: Drug: Capivasertib

INTERVENTIONS:
Drug: Capivasertib — Capivasertib will be administered orally
  Other Names: AZD5363

SUMMARY:
The purpose of this study is to measure the pharmacokinetics (PK), safety, and tolerability of capivasertib in participants with moderate hepatic impairment and participants with normal hepatic function (as control).

DETAILED DESCRIPTION:
This is a single dose, non-randomized, open-label, parallel group study. A Screening Period (Day -21 to -2): Participants in moderate impairment group will have an additional assessment of hepatic function stability on Day -7.

Treatment and Residential Period: Participants will be resident at the Investigative Site from Day -1 to Day 4 and will receive a single oral dose of capivasertib on Day 1.

Follow-up Period: Participants will return for a follow-up visit on Days 9 to 11.

ELIGIBILITY:
Key Inclusion Criteria:

* Body weight of at least 50 kg and Body Mass Index (BMI) of between ≥ 18 up to ≤ 40 kg/m2.
* Contraceptive use by participants or participant partners should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Participants must have suitable veins for cannulation or repeated venipuncture.
* Non-smoker, defined as a participant who has not smoked previously or who has discontinued smoking or the use of other nicotine/nicotine-containing products at least 3 months before the Screening Visit.
* Supporting documents confirming the participant's hepatic impairment must be available (a liver biopsy is preferable but not mandatory); participants must be classified by the Investigator as Child Pugh class B.
* Participants must meet National Cancer Institute - Organ Dysfunction Working Group (NCI-ODWG) classification of total bilirubin 1.5 to 3*upper limit of normal (ULN) and any Aspartate aminotransferase/transaminase (AST) for moderate hepatic impairment.
* Stable hepatic impairment
* For participants with normal hepatic function, Bilirubin < 1.5 × ULN, alanine aminotransferase (ALT), AST, albumin, alkaline phosphatase (ALP), gamma glutamyl transferase (GGT) < 1.2 × ULN. Creatinine < ULN. White blood cell count > lower limit of normal (LLN).

Key Exclusion Criteria:

* Any evidence of diseases (such as severe or uncontrolled systemic diseases, including uncontrolled hypertension, significant aneurysm, renal transplant and active bleeding diseases) which makes it undesirable for the participant to participate in the study or that would jeopardize compliance with the protocol.
* Refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of capivasertib.
* History of primary malignancy except for malignancy treated with curative intent with no known active disease ≥ 2 years before the first dose of study intervention and of low potential risk for recurrence. Exceptions include adequately resected non-melanoma skin cancer and curatively treated in situ disease.
* Active tuberculosis infection.
* Known Human Immunodeficiency Virus (HIV) infection, active hepatitis B or C infection, positive hepatitis C antibody, and/or positive hepatitis B virus surface antigen.
* Clinically significant abnormalities of glucose metabolism as defined by HemoglobinA1c (HbA1c) ≥ 8.0% (63.9 mmol/mol) at screening.
* Moderate or severe renal dysfunction according to age-related creatinine clearance estimated using CKD-EPI formula (i.e., creatinine clearance less than 60 mL/min).
* Fluctuating or rapidly deteriorating hepatic function.
* Presence of a hepatocellular carcinoma or acute liver disease caused by an infection or drug toxicity.
* Severe portal hypertension or surgical porto-systemic shunts.
* Biliary obstruction or other causes of hepatic impairment not related to parenchymal disorder and/or disease of the liver.
* Clinically relevant hepatic encephalopathy (Grade 3 or more).
* Severe ascites.
* Esophageal variceal bleeding (unless banded) within the past 2 months.
* Post-liver transplantation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Area under concentration time curve from zero to infinity (AUCinf) | From Day 1 to Day 4
  To compare the PK (AUCinf) of a single oral dose of capivasertib in participants with moderate hepatic impairment to participants with normal hepatic function.
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) | From Day 1 to Day 4
  To compare the PK (AUClast) of a single oral dose of capivasertib in participants with moderate hepatic impairment to participants with normal hepatic function.
Maximum plasma drug concentration (Cmax) | From Day 1 to Day 4
  To compare the PK (Cmax) of a single oral dose of capivasertib in participants with moderate hepatic impairment to participants with normal hepatic function.

SECONDARY OUTCOMES:
Concentration of capivasertib in plasma over time | From Day 1 to Day 4
  To compare the plasma concentration of a single oral dose of capivasertib in participants with moderate hepatic impairment to participants with normal hepatic function.
Area under the plasma concentration-time curve from zero to the time of the last quantifiable concentration (AUC0-t) | From Day 1 to Day 4
  To compare the PK (AUC0-t) of a single oral dose of capivasertib in participants with moderate hepatic impairment to participants with normal hepatic function.
Time to Cmax (tmax) | From Day 1 to Day 4
  To compare the PK (tmax) of a single oral dose of capivasertib in participants with moderate hepatic impairment to participants with normal hepatic function.
Terminal half-life (t½) | From Day 1 to Day 4
  To compare the PK (t½) of a single oral dose of capivasertib in participants with moderate hepatic impairment to participants with normal hepatic function.
Apparent plasma clearance (CL/F) | From Day 1 to Day 4
  To compare the PK (CL/F) of a single oral dose of capivasertib in participants with moderate hepatic impairment to participants with normal hepatic function.
Renal Clearance (CLR) | From Day 1 to Day 3
  To compare the PK (CLR) of a single oral dose of capivasertib in participants with moderate hepatic impairment to participants with normal hepatic function.
Apparent volume of distribution (Vz/F) | From Day 1 to Day 4
  To compare the PK (Vz/F) of a single oral dose of capivasertib in participants with moderate hepatic impairment to participants with normal hepatic function.
Number of participants with Adverse Events (AEs) and Serious AEs | Up to Day 11
  To examine the safety and tolerability of a single oral dose of capivasertib in participants with moderate hepatic impairment and in those with normal hepatic function.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Rialto, California
  - Research Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/